CLINICAL TRIAL: NCT04842565
Title: Phase II Trial of cTACE Plus Sintilimab for Treatment of Unresectable Intermediate-stage HCC With Beyond Up-to-seven Criteria
Brief Title: cTACE Plus Sintilimab for Unresectable Intermediate-stage HCC With Beyond Up-to-seven Criteria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, zheng wang, Associate professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-178R
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE+Sintilimab (Experimental)
  Interventions: Drug: Sintilimab; Device: TACE

INTERVENTIONS:
Drug: Sintilimab — Sintilimab (200mg ivdrip D1 Q3W)
Device: TACE — TACE will be performed by clinical demand, the interval between two TACEs is not less than 4 weeks.

SUMMARY:
This study will evaluate the efficacy and safety of Sintilimab plus Transcatheter arterial chemoembolization (TACE) in participants with Intermediate-stage unresectable hepatocellular carcinoma with Beyond Up-to-seven Criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥20 and ≤75 years old
2. Clinically diagnosed or pathologically confirmed advanced hepatocellular carcinoma. ( Fibrolamellae and mixed hepatocellular/cholangiocarcinoma subtypes are not included)
3. CNLC stage IIa/IIb or BCLC stage B, not eligible for resection or local ablation, beyond up-to-seven criteria (hepatocellular carcinomas with seven as the sum of the size of the largest tumor [in cm] and the number of tumors)
4. Newly diagnosed or recurrent more than half a year after radical surgery
5. No prior TACE treatment,
6. Child-Pugh A, ECOG PS: 0-1
7. Patients with chronic HBV infection must have HBV DNA viral load < 500 IU/mL at screening. In addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy.
8. At least one measurable site of disease as defined by modified RECIST (mRECIST) and RECICL criteria with spiral CT scan or MRI.
9. Life expectancy of at least 3 months.
10. Adequate blood count, liver-enzymes, and renal function: Haemoglobin ≥ 8.5 g/dL, absolute neutrophil count ≥ 1,500/L, platelets ≥70 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula )
11. Patients are willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.
12. Normal T3 and T4. (T3 and T4 controlled in the normal range through treatment is also eligible.)
13. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.

Exclusion Criteria:

1. Diffuse HCC or presence of vascular invasion or extrahepatic spread.
2. The patient suffered from other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ).
3. Known history of hepatic encephalopathy within 6 months
4. Known history of cardiac disease within 12 months before the first dose of study drug.
5. Clinically significant hemoptysis or tumor bleeding of any reason within 2 weeks before the first dose of study drug.
6. Severe unhealed wounds, ulcers, or fractures
7. Prior systemic anti-cancer therapy.
8. Prior treatment with TACE.
9. Suffer from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
10. Any active autoimmune disease or a history of autoimmune disease.
11. Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
12. History of allogeneic tissue/solid organ transplant.
13. Urine routine test showed urine protein ≥ ++ and confirmed 24-hour urine protein content> 1.0 g.
14. Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
15. Female patients who are pregnant, breast-feeding.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival time (mPFS) (mRECIST) | Up to approximately 24 months
  The progression-free survival time (mPFS) is defined as the date from the first TACE to the date of first documented disease progression as assessed by mRECIST or death.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 24 months
  Overall survival (OS) after enrollment is defined as the first TACE to death from any cause.
Percentage of Participants With Adverse Events | Up to approximately 24 months
  Number of participants with treatment-related adverse events as assessed by CTCAE V5.0
Objective response rate (ORR) by RECIST 1.1 and mRECIST | Up to approximately 24 months
  Objective Response Rate according to mRECIST and RECIST 1.1 for HCC
Progression-free survival time (mPFS) (RECICL) | Up to approximately 24 months
  The progression-free survival time (mPFS) is defined as the first time TACE to the date of first documented disease progression as assessed by RECICL or death, whichever comes earlier.
Time to Progression (TTP) | Up to approximately 24 months
  Time to Progression (TTP) is defined as the time from first TACE to the date of the first documented tumor progression according to the definition above.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Li L, Xu X, Wang W, Huang P, Yu L, Ren Z, Fan J, Zhou J, Zhang L, Wang Z. Safety and efficacy of PD-1 inhibitor (sintilimab) combined with transarterial chemoembolization as the initial treatment in patients with intermediate-stage hepatocellular carcinoma beyond up-to-seven criteria. J Immunother Cancer. 2025 Jan 16;13(1):e010035. doi: 10.1136/jitc-2024-010035. PMID 39824532